CLINICAL TRIAL: NCT05516823
Title: Personality and Drug Use
Acronym: PDU
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Psychedelic Data Society (Other)
Collaborators: Maastricht University (Other); Quantified Citizen Technologies Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: 21017 Personality and Drug Use
Record Dates: First submitted 2022-07-18; First posted 2022-08-26 (Actual); Last update posted 2022-09-28 (Actual); Status verified 2022-08

CONDITIONS: No Conditions Study Focus on Substance Use and Personality
Keywords: personality; substance use; psychedelics; drugs
MeSH Terms: conditions — Substance-Related Disorders

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (6):
- Group: Psychedelics-only Group: A group of participants who reported using in their past psychedelic substances only (both classical and non-classical psychedelics are included). Specifically, in the current study this group included reports on the following substances:
  Psilocybin (magic mushrooms, truffles) LSD (acid) Mescaline (peyote, San Pedro) Dimethyltryptamine (DMT) Ayahuasca 5-MeO-DMT 3-MMC Ibogaine Salvia Phenethylamines (2C family)
  Interventions: Other: Usage of drugs
- Group: Stimulants-only Group: A group of participants who reported using in their past drugs identified as stimulating compounds only (both recreational and prescribed usages are included). Stimulating compounds are considered, in the context of the current study, substances that increase the overall activity of the central nervous system. Specifically, in the current study this group included reports on the following substances:
  Cocaine Crack Amphetamines Methamphetamines Prescription stimulants (e.g., Adderall, Ritalin, Concerta)
  Interventions: Other: Usage of drugs
- Depressants-only Group: A group of participants who reported using in their past drugs identified as depressing compounds only (both recreational and prescribed usages are included). Depressing compounds are considered, in the context of the current study, substances that decrease the overall activity of the central nervous system. Specifically, in the current study this group included reports on the following substances:
  Benzodiazepines Opiates (recreational use of heroin, opium, hydrocodone, oxycodone, oxymorphone, codeine, fentanyl) Prescription opioids
  Interventions: Other: Usage of drugs
- Cannabinoids Group: A group of participants who reported using in their past cannabinoids compounds only (both recreational and prescribed usages are included). Specifically, in the current study this group included reports on the following substances:
  THC (cannabis, marijuana) CBD Medical Cannabis (both THC and CBD)
  Interventions: Other: Usage of drugs
- Psychedelic and Non-psychedelic Substances Group: A group of participants who reported using in their past drugs identified as psychedelics and stimulants and/or depressants (both recreational and prescribed usages are included). In this group participants will be included who reported using at least one non-psychedelic drug additionally to a psychedelic one. Specifically, the following options were provided:
  Psychedelic compounds:
  Psilocybin (magic mushrooms, truffles) LSD (acid) Mescaline (peyote, San Pedro) Dimethyltryptamine (DMT) Ayahuasca 5-MeO-DMT 3-MMC Ibogaine Salvia Phenethylamines (2C family)
  Non-psychedelic compounds:
  THC (cannabis, marijuana) CBD Medical Cannabis (both THC and CBD) MDMA (ecstasy) Ketamine Cocaine Crack Amphetamines Methamphetamines Prescription stimulants (e.g., Adderall, Ritalin, Concerta) Benzodiazepines Opiates (e.g., heroin, opium, hydrocodone, oxycodone, oxymorphone, codeine, fentanyl) Prescription opioids
  Interventions: Other: Usage of drugs
- Substance-naive Group: A group of participants who reported no past experience with any of the substances listed in the current study nor reported using other substances (excluding alcohol and nicotine). Participants will be assigned to this group if and only if they choose the "None of the above" option from the Substance Use Survey (item 1).

INTERVENTIONS:
Other: Usage of drugs — Self-reported past usage of drugs belonging to different chemical groups.
  Groups: Cannabinoids Group; Depressants-only Group; Group: Psychedelics-only Group; Group: Stimulants-only Group; Psychedelic and Non-psychedelic Substances Group

SUMMARY:
This is an observational, naturalistic study that aims to assess whether people with different histories of recreational or therapeutic illicit substance use (or no history at all) will differ in terms of their personalities.

DETAILED DESCRIPTION:
The study aims to assess the association between the use of various substances (including psychedelic and non-psychedelic drugs) and personality profiles. Specifically, the study will investigate if people with different histories of drug use differ in personality profiles. As psychedelics were found to influence changes in personality over time, the investigators sought to measure both the current personality profile (via the Big Five Inventory-44 (BFI)) and perceived retrospective changes in personality (via a self-constructed Retrospective Personality Scale (RPS). To investigators' knowledge, no study has explored the diversity of substance use histories in relation to individual current and retrospective personality traits and aggregate personality profiles.

The investigators aim to survey a large number of participants from all around the world, using a mobile app-based survey. The remote character of the study will increase its accessibility and diversity, which are common shortcomings in the psychedelic line of research. Additionally, a remote and anonymous study setup with no face-to-face interactions might help overcome any potential concerns participants may have regarding the sharing of sensitive information (e.g., reports on illicit substance use). To increase scientific transparency and for educational purposes (comparing personalized results with the aggregated results of participants with similar socio-demographic profiles), investigators plan to share personalized results summaries with participants of the study, which might be an additional motivating factor for study completion. In conclusion, this large-scale, low-budget, naturalistic, retrospective, observational study aims to shed light on the aforementioned gap in the literature and lay a foundation of evidence for further research.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* full legal and mental capacity
* access to a smartphone with internet to fill in the study measures (available for iOS and Android)

Exclusion Criteria:

* lack of proficiency in English
* visual impairments (not able to use mobile devices)
* illiteracy

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Adults (age of 18 or above) of full mental and legal capacities.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2022-11 (Estimated); Primary Completion 2023-11 (Estimated); Study Completion 2023-11 (Estimated)

PRIMARY OUTCOMES:
Change in scores on Big Five Inventory (BFI-44) | Measured twice: once referring to participants' personality from a period of their youth (18-21 years old) and the second time: the current moment, how they perceived their personality in general terms.
  The study will collect measures of past (youth) and current BFI scores. A separate score will be reported for each of the 5 personality traits measured by the inventory. Each score is computed by averaging the items associated with a given domain. Scores for each domain vary from 1 to 5, with higher scores meaning that a given trait is more present and noticeable in personality of the person that provided the answers.

SECONDARY OUTCOMES:
Change in scores on Retrospective Personality Scale (RPS) | Measured twice: once referring to participants' personality from a period of their youth (18-21 years old) and the second time: the current moment, how they perceived their personality in general terms.
  The study will collect measures of past (youth) and current RPS scores. A separate score will be reported for each of the 2 personality domains: positive and negative. Each of the 20 items is scored on a 3-point scale, using the following encoding: -1 (=Less), (=Without change), 1 (=More). Mean scores of 10 items for each of the domains (positive and negative) form the total score. Score Interpretation: For the positive domain, the mean score of 0 indicates no changes in personality, whereas the positive mean score (larger than 0) indicates positive changes in personality and scores below 0 point out negative changes. The reverse interpretation is true for the negative domain, with a mean score of 0 indicating no changes.

CONTACTS AND LOCATIONS:
Overall Officials: Kim PC Kuypers, PhD, Principal Investigator — Maastricht University

IPD SHARING:
Plan to Share IPD: Yes
The study will be pre-registered on the Open Science platform, where study details will be shared and regularly updated. This will be an open access project, meaning that all collected data and data analysis will be made available for all interested parties (via OSF platform). Additionally, we will share the individual summary reports with all participants who completed the study. The report will be accessible via a mobile app used to collect the study data.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: The raw data and clinical study report will be made available within 12 months from the end date of data collection.
Access Criteria: Open access
URL: https://osf.io/r3sut